CLINICAL TRIAL: NCT05983731
Title: A Pilot Observational Study to Assess the Ability of Continuous 'Home' EEG to Accurately Diagnose Narcolepsy and Demonstrate Response to Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 321547
Record Dates: First submitted 2023-07-17; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Narcolepsy Type 1; Hypersomnia
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pilot observational study is to assess the ability of continuous 'home' EEG to accurately diagnose Narcolepsy in children and young people with hypersomnia. The main question[s]it aims to answer are:

* can ambulatory home monitoring using a Dreem headband with a 'life as usual' unrestricted protocol allow accurate diagnosis of Narcolepsy, compared to gold standard in-patient PSG and MSLT
* which EEG derived sleep parameters and study duration yield most diagnostic accuracy

Participants undergoing investigation for hypersomnia will additionally be asked to wear a Dream Headband at night for weeknights, then continuously for 48 hours over the weekend. The data from the headband will then be analysed to see if it can predict the results of the polysomnography and MSLT that form routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Participants already under investigation within GSTT children and adult sleep service for hypersomnolence
* Age 12 to 25 years of age at recruitment
* Participants able to understand patient information (information including DH instructions written only in English for this initial observational study) and who can provide written informed consent or assent.

Exclusion Criteria:

* Any physician diagnosed sleep disorder (e.g. sleep apnea)
* Any physician diagnosed medical or psychiatric disorder that could explain their excessive daytime sleepiness
* Regular use of either prescribed or recreational medication that affects sleep
* Participation in another concurrent research study

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will comprise children and young adults seen in the hypersomnia clinics of the LifeSpan sleep service at Guys and St Thomas' Hospital and The Evelina London Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of diagnosis of Narcolepsy Type 1 derived by Dreem Headband compared to standard ICSD-3 protocol | 2 years
  Sensitivity (%) of Dreem headband derived EEG in predicting a final diagnosis of Narcolepsy derived from gold standard in-patient clinical testing with polysomnography and multiple sleep latency test ICSD-3 protocol.
Specificity of diagnosis of Narcolepsy Type 1 derived by Dreem Headband compared to standard ICSD-3 protocol | 2 years
  Specificity (%) of Dreem headband derived EEG in predicting a final diagnosis of Narcolepsy derived from gold standard in-patient clinical testing with polysomnography and multiple sleep latency test ICSD-3 protocol.
Positive predictive value of diagnosis of Narcolepsy Type 1 derived by Dreem Headband compared to standard ICSD-3 protocol | 2 years
  Positive predictive value (%) of Dreem headband derived EEG in predicting a final diagnosis of Narcolepsy derived from gold standard in-patient clinical testing with polysomnography and multiple sleep latency test ICSD-3 protocol.
Negative predictive value of diagnosis of Narcolepsy Type 1 derived by Dreem Headband compared to standard ICSD-3 protocol | 2 years
  Negative predictive value (%) of Dreem headband derived EEG in predicting a final diagnosis of Narcolepsy derived from gold standard in-patient clinical testing with polysomnography and multiple sleep latency test ICSD-3 protocol.

IPD SHARING:
Plan to Share IPD: No